CLINICAL TRIAL: NCT02634047
Title: Use of McGrath Videolaryngoscope to Assist Transesophageal Echocardiography Probe Insertion in Intubated Patients: A Prospective Randomized Controlled Trial
Brief Title: Use of McGrath Videolaryngoscope to Assist Transesophageal Echocardiography Probe Insertion in Intubated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH 009
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Other Complications of Surgical and Medical Procedures
Keywords: transesophageal echocardiography; videolaryngoscope; oropharyngeal injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional technique (Active Comparator): transesophageal echocardiography probe was inserted using a traditional blind insertion technique.
  Interventions: Device: conventional technique
- videolaryngoscope technique (Experimental): transesophageal echocardiography probe was advanced into esophagus under direct vision using videolaryngoscope
  Interventions: Device: videolaryngoscope technique

INTERVENTIONS:
Device: conventional technique — transesophageal echocardiography probe was inserted using a traditional blind insertion technique.
  Arms: conventional technique
Device: videolaryngoscope technique — transesophageal echocardiography probe was advanced into esophagus under direct vision using videolaryngoscope
  Arms: videolaryngoscope technique

SUMMARY:
The primary aim of this study is to investigate the difference in the first attempt and overall success rate of different techniques for insertion of transesophageal echocardiography. Secondary aim is to investigate the difference of the duration of insertion using the selected technique, complications during insertion such as oropharyngeal mucosal injury and hematoma.

DETAILED DESCRIPTION:
Eighty adult patients, who received general anaesthesia for elective open heart surgeries that required transesophageal echocardiography insertion, will be randomized by means of a computer-generated randomization order into two groups: Conventional group (Group C), and videolaryngoscope group (group VL).

Success rate of the selected technique (first attempt and overall), duration of insertion for selected technique, complications such as oropharyngeal mucosal injury and hematoma will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received general anaesthesia for open heart surgeries that required transesophageal echocardiography probe insertion

Exclusion Criteria:

* patients younger than 18 years and older than 70 years
* oropharengeal infection
* esophageal injury and anatomic abnormalities
* known or predicted difficult airway

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
difference in the first attempt and overall success rate | participants will be followed from the beginning of the transesophageal echocardiography probe insertion through the mouth to the confirmation of successful insertion (10 minutes)
  investigate the difference in the first attempt and overall success rate (with percentage) of different techniques for insertion of transesophageal echocardiography probe.

SECONDARY OUTCOMES:
difference of the duration of insertion and complications during insertion | participants will be followed for the duration of intraoperative period and postoperative 8 hours.
  investigate the difference of the duration of insertion (in seconds) using the selected technique and complications (with number and percentage) during insertion such as oropharyngeal mucosal injury and hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Nılgun Kavrut Ozturk, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Chang JE, Min SW, Kim CS, Lee JM, No H, Hwang JY. Effect of Jaw Thrust on Transesophageal Echocardiography Probe Insertion and Concomitant Oropharyngeal Injury. J Cardiothorac Vasc Anesth. 2015 Oct;29(5):1266-71. doi: 10.1053/j.jvca.2015.02.003. Epub 2015 Feb 7. PMID 25976603
- [Background] Na S, Kim CS, Kim JY, Cho JS, Kim KJ. Rigid laryngoscope-assisted insertion of transesophageal echocardiography probe reduces oropharyngeal mucosal injury in anesthetized patients. Anesthesiology. 2009 Jan;110(1):38-40. doi: 10.1097/ALN.0b013e318190b56e. PMID 19104168
- [Background] Aviv JE, Di Tullio MR, Homma S, Storper IS, Zschommler A, Ma G, Petkova E, Murphy M, Desloge R, Shaw G, Benjamin S, Corwin S. Hypopharyngeal perforation near-miss during transesophageal echocardiography. Laryngoscope. 2004 May;114(5):821-6. doi: 10.1097/00005537-200405000-00006. PMID 15126737
- [Background] Hirabayashi Y, Okada O, Seo N. Airtraq laryngoscope for the insertion of a transesophageal echocardiography probe. J Cardiothorac Vasc Anesth. 2008 Apr;22(2):331-2. doi: 10.1053/j.jvca.2007.06.012. Epub 2007 Aug 22. No abstract available. PMID 18375345
- [Background] Hirabayashi Y. GlideScope-assisted insertion of a transesophageal echocardiography probe. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):628. doi: 10.1053/j.jvca.2006.11.015. Epub 2007 Feb 22. No abstract available. PMID 17678807